CLINICAL TRIAL: NCT01814449
Title: Department of Breast Surgery And Department of Nuclear Medicine, Fudan University Shanghai Cancer Center,
Brief Title: Relationship Between Hypoxia and Endocrine Response in Human Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guangyu Liu, Deputy director of Department of Breast Surgery,Cancer Hopital & Institute, Fudan University
Other Study IDs: 20120224.1.1
Record Dates: First submitted 2013-03-16; First posted 2013-03-20 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer; Hypoxia
Keywords: Breast cancer; Hypoxia; Hypoxia related gene; Endocrine therapy; Treatment resistance
MeSH Terms: conditions — Breast Neoplasms; Hypoxia | interventions — Letrozole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Each patient underwent diagnostic core-needle biopsy on the primary site at baseline. A therapeutic surgery or a second core-needle biopsy on the primary site was planned in a subset of patients after at least 3 months of primary letrozole therapy. Both biopsy and surgical samples of primary tumors were routinely embedded in paraffin wax and cut to 3- to 5-mm thickness and dried overnight for immunohistochemistry testing.Immunohistochemistry staining for HIF-1-alpha and Ki67 were performed on 3- to 5-mm serial sections on coated slides.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hypoxic Group: Higher 18FMISO uptake (Target to background Ratio, TBR>1.2) in Primary breast cancer by 18FMISO PET/CT scan.Primary endocrine therapy Letrozole was given to the patients.
  Interventions: Other: 18FMISO PET/CT scan; Drug: Letrozole
- Non-Hypoxic Group: Lower 18FMISO uptake (TBR<1.2)in primary breast cancer by 18FMISO PET/CT scan.Primary endocrine therapy letrozole was given to the patients.
  Interventions: Other: 18FMISO PET/CT scan; Drug: Letrozole

INTERVENTIONS:
Other: 18FMISO PET/CT scan — The baseline 18F-FMISO PET/CT scans were scheduled before initiation of endocrine therapy. All patients were injected intravenously with 370 MBq of 18F-FMISO and PET/CT static emission scans were conducted at 4 hours after injection.
Drug: Letrozole — Patients were assigned to primary endocrine therapy with letrozole 2.5mg daily for at least 4 months.

SUMMARY:
The aim of our current study was to analyze whether 18F-labeled Fluoromisonidazole (1-(2-nitro-1-imidazolyl)- 2-hydroxy-3-fluoropropane [18F-FMISO]) PET/CT and expression of HIF-1-alpha could predict response of primary endocrine therapy in ER-positive breast cancer

DETAILED DESCRIPTION:
Approximately 30% of ER-positive breast cancer will unfortunately display primary resistance to hormonal therapy, and some may develop acquired resistance to the therapy after initial treatment. Hypoxia is a normal phenomenon in solid tumors that arises, in part, from uncontrolled proliferation and immature blood vessels. Previous studies have demonstrated hypoxia significantly reduced both the growth-promoting effects of estradiol (E2) and the growth-inhibitory effects of an antiestrogen on ER-positive breast cancer cell lines. A recent study comparing neoadjuvant letrozole with letrozole plus metronomic cyclophosphamide found that increased levels of HIF-1a were significantly associated with resistance to treatment. Taken together, these data indicate that hypoxia might be associated with endocrine resistance in breast cancer.

With PET/CT, radiolabeled hypoxia-avid compounds can be applied to evaluate oxygenation status in experimental or human tumors. 18F-labeled fluoromisonidazole (1-[2-nitro- 1-imidazolyl]-2-hydroxy-3-fluoropropane [18F-FMISO]) PET/CT is the most widely used one in the clinic. Studies have demonstrated an excellent correlation between the 18F-FMISO uptake and oxygenation status of several cancers including breast cancer.

The major aim of our study was to analyze uptake of 18FFMISO as well as the IHC expression of HIF-1-alpha in ER-positive breast cancers, and to predict the clinical, pathological and biological response of primary endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal female
2. With primary invasive ER positive breast cancer pathologically approved by core needle biopsy
3. The target lesion must be measurable and maximum diameter should be over 2cm.
4. Require and accept Endocrine therapy
5. Never treated with endocrine therapy before
6. Patients must have an ECOG performance status of 0 to 2
7. Leucocyte count must be ≥ 3.0*10^9/L and platelet count must be ≥ 40*10^9/L; AST/SGOT or ALT/AGPT must be < 2 times the ULN; serum creatinine must be < 2 times the ULN

Exclusion Criteria:

1. Patients with brain and liver metastasis
2. Previous history of severe heart dysfunction (above Class III), infection, osteoporosis, bone related event or disease in endocrine system
3. Combination of other anticancer therapy, with the exception of biphosphonate

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women who had ER-a-positive breast cancer at stages II-IV and had never received prior endocrine therapy were considered eligible for this study.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-02 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Clinical Objective Response | 4 months
  Tumor response was evaluated according to the criteria of the World Health Organization. Clinical tumor progression (PD) was defined as an increase of at least 25% in tumor size; stable disease (SD) as an increase of less than 25% or a reduction of less than 50%; partial response (cPR) as a tumor shrinkage greater than 50%; and complete response (cCR) as the complete disappearance of all clinical signs of disease.

SECONDARY OUTCOMES:
Pathological Response | 4 months
  Including pathological complete response (pCR or Grade 5),pathological partial response (pPR or Grade 3-4) and pathological non-response (NR or Grade 1-2).
Depression of Ki67 score | 3 months
  A biological response of Ki67 depression was tested on a second core needly biopsy on the primary site of the breast cancer after 3 months of primary endocrine therapy. Ki67>=15% was regarded as a biological resistance to primary endocrine therapy

OTHER OUTCOMES:
Disease free survival | 5 years
  An early recurrence of the disease during adjuvant endocrine therapy was also regarded as a resistance to endocrine therapy

CONTACTS AND LOCATIONS:
Overall Officials: Guangyu Liu, M.D., Principal Investigator — Cancer Hospital/Institute,Fudan University
Locations (1):
- Cancer Hospital/ Institute, Fudan University, Shanghai, Shanghai Municipality, China